CLINICAL TRIAL: NCT04962347
Title: Real World Study of COVID-19 in a Flyover Region
Status: Completed | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-112
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: Remdesivir
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Real world data are needed on remdesivir (RDV) efficacy in COVID-19, especially in the underserved populations of the United States (U.S.) Gulf Coast as initial clinical trials may not be representative of this population. Specifically, regions such as New Orleans are 60% African American, a much greater proportion of African Americans than initial RDV studies. The main hypothesis is that a real world data based study will provide specific information related to RDV efficacy in COVID-19 patients from underserved / underrepresented populations of the U.S. Gulf Coast. The main goal of this study is to provide population-centered information related on RDV related to indication (stage of disease), dosing, monitoring, efficacy and contraindications for future COVID-19 patients in this underserved region.

DETAILED DESCRIPTION:
This study involves extracting data from 10,000 patients with Polymerase Chain Reaction (qPCR) confirmed COVID-19 infection through electronic-charts of Tulane Medical Center and University Medical Center (New Orleans, Louisiana) and Doctors Hospital at Renaissance (DHR) system (Texas). According to the inclusion criteria below and spanning from September 2019 - December 2021 we predict to include 1500 RDV treated patients and 8500 non-treated comparators, all with COVID-19, through the Research Action for Health Network (REACHnet) (link: https://eco.reachnet.org) in partnership with the Louisiana Public Health Institute (LPHI).

Statistical plan:

Following anonymized data extraction, propensity score will be used to compare primary and secondary endpoints between matched COVID-19 infected patients who received RDV to those who did not receive RDV. Patients of both cohorts will be stratified by severity. Moderate and severe respiratory distress associated with COVID-19 are defined as per US-GS-540-5773 and US-GS-540-5774 clinical trials. Through the investigator's extensive Electronic Medical Record (EMR) data collection network including diverse underserved populations of the U.S. Gulf South, they will evaluate real world outcomes of RDV treatment for COVID-19. The 2 cohorts will be compared with focus upon respiratory distress evolution, co-morbidities and other illness associated/relevant to COVID-19 course during admission, post-discharge during convalescent period of up to 6 months, and documentation of pre-admission comorbidities in the 6 months pre-admit.

ELIGIBILITY:
Inclusion Criteria:

* Positive qRT PCR for COVID-19 from a nasopharyngeal, nasal, or oropharyngeal swab or from bronchoalveolar lavage.
* Received RDV (cases) or did not receive RDV (controls).
* Age ≥ 18 years

Exclusion Criteria:

- None.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 infected patients who received remdesivir to be compared to those who did not receive remdesivir.
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
The change of clinical severity, as measured using 7-point ordinal clinical severity scale, from first RDV dose through day 11 post-dose. | Change from Day 1 to Day 11
  Clinical severity will be measured using 7-point ordinal scale (1 Death, 2 Hospitalized, on invasive mechanical ventilation or Extracorporeal membrane oxygenation (ECMO), 3 Hospitalized, on non-invasive ventilation or high flow oxygen devices, 4 Hospitalized, requiring low flow supplemental oxygen (less than 15L), 5 Hospitalized, not requiring supplemental oxygen-requiring ongoing medical care (COVID-19 related or otherwise), 6 Hospitalized, not requiring oxygen-no longer requires ongoing medical care, 7 Not hospitalized. The improvement and change in clinical severity, from first RDV dose recorded as Day 1 to Day 11 is recorded.

SECONDARY OUTCOMES:
Mortality during admission | 6 months
  Mortality rate change during admission compared between RDV vs non-RDV subjects
Mortality at 6 months following symptom onset | 6 months
  Mortality rate through end of study period (6 months following symptom onset) compared between RDV vs non-RDV subjects
Post-COVID-19 symptoms | 6 months
  Impact measurement of acute COVID-19 RDV on post-COVID-19 symptoms/morbidity compared between RDV vs non-RDV subjects
Post-COVID-19 mortality | 6 months
  Impact measurement of acute COVID-19 RDV on post-COVID-19 mortality compared between RDV vs non-RDV subjects

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Drouin, MD, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States